CLINICAL TRIAL: NCT02286323
Title: Can the Bonfils Intubation Fiberscope Rival the Macintosh Laryngoscope During Resuscitation With Uninterrupted Chest Compression?
Brief Title: Endotracheal Intubation During Resuscitation
Acronym: EIDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/07
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: Intubation, Endotracheal
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endotracheal intubation without chest compressions (Experimental): Endotracheal intubation of mannikin during resuscitation without chest compressions.
  Interventions: Device: Bonfils; Device: Macintosh
- Endotracheal intubation with uninterrupted chest compressions (Experimental): Endotracheal intubation of mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: Bonfils; Device: Macintosh

INTERVENTIONS:
Device: Bonfils — Bonfils Intubation Fiberoscope
Device: Macintosh — Direct laryngoscopy using Macintosh Laryngoscope

SUMMARY:
We hypothesized that the BONFILS is beneficial for intubation of manikins while performing CPR. In the current study we compared the performance of the BONFILS and the Macintosh laryngoscopes with respect to their effectiveness and time to successful ETI during chest compression (CC) using an adult manikin.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (paramedics, nurses, physicians)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | intraoperative
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | intraoperative
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
POGO score | 1 day
  self-reported percentage of glottis opening (POGO) score

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Kurowski, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland